CLINICAL TRIAL: NCT05933811
Title: Does the Contralateral Testicular Volume Decide the Need for Diagnostic Laparoscopy in Cases of Unilateral Impalpable Undescended Testis?
Brief Title: Contralateral Testicular Volume in Unilateral Impalpable Testis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Principal Investigator, Ahmed Elrouby, Associate Professor of pediatric Surgery, Egyptian Biomedical Research Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0305079
Record Dates: First submitted 2023-05-26; First posted 2023-07-06 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Pediatric ALL
Keywords: Impalpable testis; volume; Ultrasound
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric patients with unilateral impalpable maldescended testis (Experimental): Patients in the pediatric age group who presented by unilateral impalpable undescended testis
  Interventions: Procedure: exploratory laparoscopy

INTERVENTIONS:
Procedure: exploratory laparoscopy — Laparoscopic exploration for impalpable maldescended testis in pediatric age group

SUMMARY:
This prospective interventional study aimed at the preoperative sonographic estimation of the testicular volume of the normal side in case of contralateral impalpable maldescended testis in order to predict the condition of the diseased side and hence the need for diagnostic laparoscopy.

DETAILED DESCRIPTION:
Purpose: This study aimed at the evaluation of the value of the estimated volume of a normal testis to predict the status of its contralateral impalpable side and hence decide the importance of laparoscopic exploration. Material & methods: Patients with unilateral impalpable maldescended testis - as confirmed by clinical and sonographic examination- were enrolled in this prospective interventional study between November 2018 and August 2022 at Elshatby University Hospital, Faculty of Medicine, Alexandria University. The volume and three-dimensional diameter of the normal contralateral testis were measured by the pre-operative US using the formula: Volume = L x W x H x π/6, where L is the length, W is the width, H is the height, and was correlated with the intra-operative laparoscopic findings.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with unilateral impalpable maldescended testis

Exclusion Criteria:

* Patients with bilateral impalpable maldescended testis and those with post-operative ascended testis

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
The size of the impalpable testis as examined by laparoscopy | Intraoperative
  The size of the testis in millimeters
The presence of testicular vessels of the impalpable testis as examined by laparoscopy | Intraoperative
  The presence or absence of testicular vessels
The presence of the vas deference of the impalpable testis as examined by laparoscopy | Intraoperative
  The presence or absence of the vas deference

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Elrouby, MD, Principal Investigator — Pediatric Surgery department
Locations (1):
- Faculty of Medicine, Alexandria, Egypt

REFERENCES:
- [Derived] Elrouby A, Ghalab M, Kotb M. Does the contralateral testicular volume decide the need for diagnostic laparoscopy in cases of unilateral impalpable undescended testis? BMC Urol. 2024 Mar 26;24(1):68. doi: 10.1186/s12894-024-01455-2. PMID 38532380

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT05933811/Prot_SAP_001.pdf